CLINICAL TRIAL: NCT03961776
Title: Monitoring Treatment Response With On-board DWI During Neo-adjuvant Chemo-radiation for Rectal Cancer Using Magnetic Resonance-guided-radiotherapy Systems
Acronym: DWI_RECT_MRGRT
Status: Recruiting | Type: Observational
Sponsor: Institut Paoli-Calmettes (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Other Study IDs: DWI_RECT_MRGRT-IPC 2019-002
Record Dates: First submitted 2019-05-20; First posted 2019-05-23 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Rectal Adenocarcinoma
Keywords: Diffusion weighted imaging; Radiation therapy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- non-metastatic rectal adenocarcinoma nRCT indicated: Patients with histologically confirmed non-metastatic rectal adenocarcinoma and for whom treatment with nRCT has been indicated.
  Interventions: Device: MRI-guided radiotherapy by on-board DWI sequences

INTERVENTIONS:
Device: MRI-guided radiotherapy by on-board DWI sequences — The radiotherapy treatment will be delivered on the MRI-guided radiotherapy platform. The on-board DWI sequences will be performed every three fractions in addition to the treatment session and will last approximately 3-4 minutes.

SUMMARY:
feasibility of using a diffusion sequence of a MRgRT system as an early marker of treatment response during nRCT of rectal adenocarcinoma.

DETAILED DESCRIPTION:
feasibility of using a diffusion sequence of a MRgRT system as an early marker of treatment response during nRCT of rectal adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Patient over 18 years old.
2. Diagnosis of histologically confirmed rectal adenocarcinoma for which nRCT has been indicated.
3. Karnofsky Index (KPS) ≥ 70 or ECOG = 0 or 1
4. Signed consent to participation.
5. For women of childbearing age, effective contraception must also be agreed for the duration of treatment.
6. Affiliation to a social security regimen, or beneficiary of such a regimen.

Exclusion Criteria:

1. Predominant mucinous component on initial MRI, biopsy and / or definitive pathology. Mucin may lead to overestimation of ADC values on DWIs.
2. Contraindications to the MRI procedure (non compatible pacemaker or other metallic foreign body, severe claustrophobia).
3. Exclusive radiation therapy.
4. Other associated neo-adjuvant treatment.
5. Delayed completion of the surgery (more than approximately 10 weeks after the end of the nRCT) or cancellation of the surgical procedure.
6. Contraindications to capecitabine: Severe hepatic impairment, severe renal impairment (creatinine clearance <30 ml / min),
7. Known deficiency of Dihydropyrimidine dehydrogenase (DPD), known hypersensitivity to 5-FU / capecitabine and / or its excipients.
8. Participation in a protocol with concurrent treatment.
9. Pregnant or likely to be pregnant (without effective contraception) or breastfeeding
10. Person in emergency situation, person of legal age subject to a legal protection measure, or unable to express his / her consent.
11. Impossibility of attending the medical examination of the test for geographical, social or psychological reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of men and / or women over 18 years of age, with no upper limit age, with histologically confirmed non-metastatic rectal adenocarcinoma and for whom treatment with nRCT has been indicated.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Estimated)
Dates: Start 2020-06-08 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Predictive value of Apparent Diffusion Coefficient measured using MRgRT system | At surgery (5 to 10 weeks after completion of chemoradiation)
  Pathological complete response using AJCC criteria

CONTACTS AND LOCATIONS:
Overall Officials: Marguerite TYRAN, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (2):
- University of California Los Angeles (UCLA), Los Angeles, California, United States
- Institut Paoli Calmettes, Marseille, Bouches Du Rhone, France

IPD SHARING:
Plan to Share IPD: No